CLINICAL TRIAL: NCT03614286
Title: Trichomonas Vaginalis Genotyping in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, nasser mohamed abdelkareem, Assistant Lecturer of Medical Parasitology, Assiut University
Other Study IDs: T V Genotyping
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Trichomonas Vaginalis Genotyping in Upper Egypt; Vaginitis Trichomonal
MeSH Terms: conditions — Trichomonas Vaginitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — vaginal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: culture and pcr — The swab immersed in Diamond's Modified medium culture tube and squeezed for cultivation and examined daily with a light microscope to identify T. vaginalis Samples from culture will be placed in 1 ml of a commercial PCR transport medium (AMPLICOR; Roche Diagnostic Systems, Branchburg, N.J.) and kept at 4°C until arrival at the laboratory within 4 days of collection. An equal volume of specimen diluent (AMPLICOR) was added to the sample , and the preparation was mixed, incubated at room temperature for 10 min, and stored at -70°C until tested.
  Other Names: PCR

SUMMARY:
The worldwide incidence of trichomoniasis was estimated to be 276.4 million new cases per year in 2008 .In Egypt, the reported prevalence rate ranges from 5% to 79.16% we aim to study genetic variability of Trichomonas vaginalis using PCR

DETAILED DESCRIPTION:
In women, trichomoniasis has a wide range of presentations, from asymptomatic to acute or chronic inflammatory disease they include urethral discharge and dysuria. Among women, common sites of infection include the vagina, urethra and endocervix. Symptoms include vaginal discharge (which is often diffuse, malodorous, yellow-green), dysuria, itching, vulvar irritation and abdominal pain. The normal vaginal pH is 4.5, but with TV infection this increases markedly, often to >5 Colpitis macularis or strawberry cervix is seen in about 5 % of women, though with colposcopy this rises to nearly 50 % .Other complications include infection of the adnexa, endometrium, and Skene and Bartholin glands. In men, it can cause epididymitis, prostatitis, and decreased sperm cell motility .

A lot of risk factors of infection are related to age, educational level, residence, race/ethnicity, marital status, number of sex partners, use of condom/IUD, history of sexually transmitted diseases and presence of vaginal discharge .

Traditionally physicians make the diagnosis based on clinical grounds, but in women, the characteristics of the vaginal discharge, including color and odor, are poor predictors of T. vaginalis. Since no symptom alone or in combination is sufficient to diagnose T. vaginalis infection reliably, laboratory diagnosis is necessary ,Diagnosis of T. vaginalis infection is established by the traditional method wet mount test, in which "corkscrew" motility observed . Anyhow, culture has long been the gold standard for diagnosing T. vaginalis infection , with a sensitivity range from 85-95 % . Other used methods for diagnosis include enzyme-linked immunosorbent assay , staining methods latex agglutination , immunochromatography and nucleic acid amplification tests .In order to develop protocol for the diagnosis of trichomoniasis, ideal test should have high sensitivity and specificity and be easily available, simple to perform, and inexpensive Knowledge of the genetic characteristics of T. vaginalis populations is valuable for the prevention and control of trichomoniasis in humans .

The lengths of specific regions in the small subunit of nuclear ribosomal RNA (SSU nrRNA, also known as 18S rRNA) are not conserved among different groups, and these differences can be significant. Thus, 18S rRNA is suitable to study genetic variations and genotypes of organisms.

The use of reliable classification and genetic characterization methods can help to clarify the ambiguities in this field.

Multiple approaches to typing Trichomonas isolates have been described; antigenic characterization, ribosomal gene and intergenic region sequence polymorphisms, random amplified polymorphic DNA analysis, and restriction fragment length polymorphism .These studies produced differing results, even when using similar techniques, in attempting to demonstrate concordance between parasite genotypes and phenotypic expressions during infection, such as virulence and metronidazole resistance. The T. vaginalis genome composition provides a potential explanation for this difficulty in correlating genotype with phenotype.

ELIGIBILITY:
Inclusion Criteria:

* females ,non virgins,complain from vaginitis ,at reproductive age and attending to sohag general hospital outpatient clinic of gynecology and obstetric

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — non virgins females
Study Population: one group from 20 patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
study genetic variability of Trichomonas vaginalis using PCR | 1year
  detection of TV in vaginal swap then PCR done to detect genetic diversity

REFERENCES:
- [Background] Zhang Z, Kang L, Wang W, Zhao X, Li Y, Xie Q, Wang S, He T, Li H, Xiao T, Chen Y, Zuo S, Kong L, Li P, Li X. Prevalence and genetic diversity of Trichomonas vaginalis clinical isolates in a targeted population in Xinxiang City, Henan Province, China. Parasit Vectors. 2018 Mar 2;11(1):124. doi: 10.1186/s13071-018-2753-4. PMID 29499747